CLINICAL TRIAL: NCT01329380
Title: Special Investigation (All Cases Investigation in Patients With Ankylosing Spondylitis)
Brief Title: Special Investigation in Patients With Ankylosing Spondylitis (All Patients Investigation)
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P12-764
Record Dates: First submitted 2011-03-17; First posted 2011-04-05 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2018-12

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adalimumab: Participants with ankylosing spondylitis (AS) receiving treatment with adalimumab (Humira) as prescribed by their physician.

SUMMARY:
This study of adalimumab (Humira) will be conducted to clarify the following with regard to the treatment of ankylosing spondylitis with this drug:

* Unknown adverse drug reactions (especially important adverse drug reactions)
* Incidence and conditions of occurrence of adverse reactions in the clinical setting
* Factors that may affect the safety and effectiveness of Humira

ELIGIBILITY:
Inclusion Criteria:

* Patients with ankylosing spondylitis who are not responding well to conventional therapy and receive adalimumab will be enrolled in the survey

Exclusion Criteria:

* Contraindications according to the Package Insert

  * Patients who have serious infections
  * Patients who have tuberculosis
  * Patients with a history of hypersensitivity to any ingredient of Humira
  * Patients who have demyelinating disease or with a history of demyelinating disease
* Patients who have congestive cardiac failure

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who receive Humira for the treatment of ankylosing spondylitis
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2010-10-27 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (194):
- Japan (194):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - Hyogo College of Medicine Hosp, Nishinomiya, Hyōgo
  - Yokohama City Univ Medical Ctr, Yokohama, Kanagawa
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka City University Hospital, Osaka, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Shiga Univ Med Science Hosp, Ōtsu, Shiga
  - Medical Hospital of Tokyo Medical and Dental University, Bunkyo-ku, Tokyo
  - St. Luke's International Hosp, Chūō, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Teikyo University Hospital, 板橋区, Tokyo
  - Asano Orthopedic Clinic, Aichi
  - Nagoya Daini Red Cross Hosp, Aichi
  - Ozone Surgery Clinic, Aichi
  - Yamagiwa Clinic, Aichi
  - Narushima Internal Med Clinic, Ami-machi
  - Katayama Orthopedic Rheum Clin, Asahikawa
  - Asahikawa Med College Hosp, JP, Asahikawa
  - Asahikawa Kosei General Hosp, Asahikawa-shi
  - Atsugi City Hospital, Atsugi-shi
  - Chiba University Hospital, Chiba
  - University of Yamanashi Hosp, Chūō
  - Tama Medical Center, Fuchū
  - Fujieda Municipal General Hosp, Fujieda
  - Nakamura Clinic, Fukuchiyama-shi
  - Hamanomachi Hospital, Fukuoka
  - NHO Kyushu Medical Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - JP Red Cross Fukuoka Hosp, Fukuoka
  - Mutaguchi Orthopedics Clinic, Fukuoka
  - PS Clinic, Fukuoka
  - Fukushima Med Univ Hosp, Fukushima
  - Fukushima Red Cross Hospital, Fukushima
  - Minami Tohoku Fukushima Hosp, Fukushima
  - Gifu University Hospital, Gifu
  - Seirei Mikatahara General Hosp, Hamamatsu
  - Osaka Rehabilitation Hospital, Hannan
  - Matsunami General Hospital, Hashima-gun
  - Kono Orthop. and Int. Med Clin, Higashimatsuyama-shi
  - Tama-Hokubu Medical Center, Higashimurayama
  - Yamaguchi Clinic, Higashiosaka-shi
  - NHO Higashi-Ohmi Gen Med Ctr, Higashiōmi
  - NHO Himeji Medical Center, Himeji
  - Hirosaki Uni School Med & Hosp, Hirosaki
  - Hirosaki Memorial Hospital, Hirosaki
  - Hiroshima Red Cross Hosp Atomi, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Yamana-kai Higashi Hiroshima, Hiroshima
  - Hiroshima Clinic, Hiroshima
  - Shigenobu Clinic, Hiroshima
  - Midori Hospital, Hyōgo
  - Kohnodai Hospital, Ichikawa-shi
  - Iwate Prefectural Iwai Hosp, Ichinoseki-shi
  - Saitama Medical University Hos, Iruma-gun
  - Suga Orthopedic Hospital, Isahaya
  - Isahaya Health Ins Genl Hosp, Isahaya
  - NHO Iwakuni Clinical Center, Iwakuni-shi
  - Juntendo Univ Shizuoka Hosp, Izunokuni-shi
  - Kaga City Hospital, Kaga-shi, Ishikawa
  - Kagoshima Red Cross Hospital, Kagoshima
  - Kagoshima Univ Medical and Den, Kagoshima
  - Kameda Medical Center, Kamogawa
  - Saiseikai Kanazawa Hospital, Kanazawa
  - Kanazawa University Ho, Kanazawa
  - Kasugai Orthopaedic Clinic, Kasugai
  - Asahi Hospital, Kasugai
  - NHO Osaka Minami Med Ctr, Kawachi-Nagano
  - Nagasawa Clinic, Kawagoe-shi
  - St. Marianna Univ Hospital, Kawasaki
  - Edakuni Orthopedic Clinic, Kiryū
  - JR Kyushu Hospital, Kitakyushu
  - Univ Occup & Environ Health, Kitakyushu
  - Kobe University Hospital, Kobe
  - Komaki Daiichi Hospital, Komaki
  - Jusendo General Hospital, Koriyama-shi
  - Juntendo Univ Koshigaya Hosp, Koshigaya
  - Saiseikai Kyoto Hospital, Kōtari
  - Shunan Memorial Hospital, Kudamatsu-shi
  - Kumamoto Rheumatology Clinic, Kumamoto
  - Kunitachi Clinic, Kunitachi
  - Kawasaki Medical School Hosp, Kurashiki
  - Kurashiki Central Hospital, Kurashiki
  - Jujo Rehabilitation Hospital, Kyoto
  - Kyoto Prefect Univ Med, Kyoto
  - JP Red Cross Kyoto Daiichi Hos, Kyoto
  - Kagawa University Hospital, Kyoto
  - Iwasaku Orthopedic Clinic, Kyoto
  - Tori Clinic, Maizuru-shi
  - Matsuyama Red Cross Hosp, Matsuyama
  - Mino Municipal Hospital, Mino
  - Suzuki Orthopedic Clinic, Miyashiro-machi
  - Miyazaki Prefectural Miyazaki, Miyazaki
  - Iwate Medical University Hosp, Morioka
  - Noguchi Seikeigeka Naika Iin, Motosu-shi
  - Munakata Medical Assoc. Hosp., Munakata-shi
  - Aichi Medical University Hosp, Nagakute
  - Chukyo Social Insurance Hospit, Nagoya
  - NHO Nagoya Medical Center, Nagoya
  - Shinseikai Daiichi Hospital, Nagoya
  - Higashi Hosp City of Nagoya, Nagoya
  - Kakinuma Orthopedics Clinic, Nagoya
  - Oura Clinic, Naha
  - Kochi Medical School Hospital, Nankoku-shi
  - Nara City Hospital, Nara
  - Asahigaoka Hospital, Nara
  - Mitsuka Rheumatism Clinic, Narashino-shi
  - Niigata City General Hospital, Niigata
  - Nirasaki City Hospital, Nirasaki
  - Nisshin Orido Hospital, Nisshin
  - Yamachika Memorial Gen Hosp, Odawara-shi
  - Ohama Daiichi Hospital, Okinawa
  - Yuri Plastic Surgery, Ono
  - Yukioka Hospital, Osaka
  - Osaka Saiseikai Noe Hospital, Osaka
  - NTT WEST Osaka Hospital, Osaka
  - Osaka Red Cross Hospital, Osaka
  - Kansai Medical Univ Takii Hosp, Osaka
  - Kojima Orthopedic Clinic, Osaka
  - Murakami Orthopaedics Clinic, Osaka
  - Osaka Rheumatology Clinic, Osaka
  - Ushio Clinic, Osaka
  - Yodogawa Christian Hospital, Osaka
  - Oita Red Cross Hospital, Ōita
  - Saiseikai Hita Hospital, Ōita
  - Sunrise Sakai Hospital, Ōita
  - Ome Municipal General Hospital, Ōme
  - Osaki Citizen Hospital, Ōsaki
  - Ota Memorial Hospital, Ōta-ku
  - Saga University Hospital, Saga
  - Osaka Rosai Hospital, Sakaishi
  - Yoshida Internal Med Clinic, Sakaki
  - Kyoto University Hospital, Sakyo-ku
  - Teine Internal Med Rheuma Clin, Sapporo
  - Teine Keijinkai Clinic, Sapporo
  - Sapporo Medical Univ Hosp, Sapporo
  - Kin-ikyo Chuo Hospital, Sapporo
  - KKR Sapporo Med Ctr Tonan Hosp, Sapporo
  - Sasebo Chuo Hospital, Sasebo
  - Sasebo City General Hospital, Sasebo-shi
  - Tohoku University Hospital, Sendai
  - NHO Nishitaga National Hospita, Sendai
  - Tohoku Pharmaceutical Univ Hos, Sendai
  - Jyunshinkai Inoue Hospital, Seto
  - Niigata Rheumatic Center, Shibata
  - Saiseikai Suita Hospital, Suita
  - Osaka University Hospital, Suita
  - Hirose Clinic, Tokorozawa
  - Kotesashi Orthopedic Clinic, Tokorozawa-shi
  - Hishita-Hiasa Neurosurgery and, Tokushima
  - Toyo Hospital, Tokushima
  - Kyoundo Hospital, Tokyo
  - Mitsui Memorial Hospital, Tokyo
  - The Jikei University Hospital, Tokyo
  - Toranomon Hospital, Tokyo
  - The University of Tokyo, Tokyo
  - Juntendo University Hospital, Tokyo
  - Tokyo Metropolitan Bokutoh Hos, Tokyo
  - Keiyo Hospital, Tokyo
  - Toho Univ Med Ctr Omori Hosp, Tokyo
  - Tokyo Medical University Hosp, Tokyo
  - National Ctr Global Health Med, Tokyo
  - Tokyo Womens Med Univ Hosp, Tokyo
  - Kawakita General Hospital, Tokyo
  - Nihon University Itabashi Hosp, Tokyo
  - Juntendo Univ Nerima Hosp, Tokyo
  - JP Red Cross Musashino Hosp, Tokyo
  - Akasaka Chuo Clinic, Tokyo
  - Edogawa Hospital, Tokyo
  - Ishigaki Orthopedic Clinic, Tokyo
  - Kanamecho Hospital, Tokyo
  - Matsuda Orthopedic Rheuma Clin, Tokyo
  - NHO Disaster Medical Center, Tokyo
  - Showa University Hospital, Tokyo
  - Yoshida Internal Med Clinic, Tokyo
  - Matsuno Clinic Rheumatic Disea, Toyama
  - Toyama Prefectural Ctr Hosp, Toyama
  - Fujita Health University Hosp, Toyoake
  - Toyama University Hospital, Toyoma
  - Toyooka Hospital, Toyooka
  - Kishi Orthopedics Medical Clin, Tsuchiura-shi
  - Tsukuba University Hospital, Tsukuba
  - Tsuyama Chuo Memorial Hospital, Tsuyama
  - Daini Okamoto General Hospital, Uji
  - Wakayama Medical University, Wakayama
  - Yamagata University Hospital, Yamagata
  - Yamagata City Hosp Saiseikai, Yamagata
  - Yamaguchi Red Cross Hospital, Yamaguchi
  - Shuto General Hospital, Yanai-shi
  - Kumamoto Rosai Hospital, Yatsushiro-shi
  - Showa Univ N Yokohama Hosp, Yokohama
  - Tottori University Hospital, Yonago-shi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four hundred and three participants were registered at 195 sites in Japan. Survey forms were available for 400 participants from 194 sites.
Period: Overall Study
Arm/Group | Adalimumab
Started (Participants who were registered) | 403
Safety Population (Excludes duplicate participants and participants starting treatment prior to study registration) | 396
Completed (Participants with available efficacy data at 12 weeks or 24 weeks after the start of treatment) | 374
Not Completed | 29

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Arm/Group | Adalimumab
Number analyzed (Participants) | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (15.6)
Age, Customized [Count of Participants; unit: Participants]
  15 to < 65 years | 344
  ≥ 65 years | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130
  Male | 266
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 396
Region of Enrollment [Number; unit: participants]
  Japan | 396

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) is an injury caused by taking a medication, in which a causative relationship can be shown.
  A serious adverse drug reaction is any untoward medical occurrence that at any dose;
  * Results in death
  * Life threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent of significant disability or incapacity
Time Frame: 24 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 396
Participants
  Adverse drug reactions | 101
  Serious adverse drug reactions | 15

2. Primary Outcome: Number of Participants With Adverse Drug Reactions by Baseline Factors
Description: An adverse drug reaction (ADR) is an injury caused by taking a medication, in which a causative relationship can be shown. ADRs are reported by baseline characteristics.
  NSAID: non-steroidal anti-inflammatory drug
  DMARD: disease-modifying anti-rheumatic drug
  BASDAI: Bath Ankylosing Spondylitis Disease Activity Index
Time Frame: 24 weeks
Population: Safety analysis set; results are only included for participants with non-missing baseline data for each characteristic.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 396
Participants
  Age: 15 to < 65 years: number analyzed (Participants) | 344
  Age: 15 to < 65 years | 94
  Age: ≥ 65 years: number analyzed (Participants) | 52
  Age: ≥ 65 years | 7
  Sex: Male: number analyzed (Participants) | 266
  Sex: Male | 66
  Sex: Female: number analyzed (Participants) | 130
  Sex: Female | 35
  Body Mass Index: < 18.5 kg/m²: number analyzed (Participants) | 31
  Body Mass Index: < 18.5 kg/m² | 9
  Body Mass Index: 18.5 - < 25 kg/m²: number analyzed (Participants) | 164
  Body Mass Index: 18.5 - < 25 kg/m² | 36
  Body Mass Index: 25 - 30 kg/m²: number analyzed (Participants) | 63
  Body Mass Index: 25 - 30 kg/m² | 25
  Body Mass Index: ≥ 30 kg/m²: number analyzed (Participants) | 25
  Body Mass Index: ≥ 30 kg/m² | 5
  Duration of illness: < 5 years: number analyzed (Participants) | 129
  Duration of illness: < 5 years | 34
  Duration of illness: 5 to < 10 years: number analyzed (Participants) | 80
  Duration of illness: 5 to < 10 years | 21
  Duration of illness: 10 to < 20 years: number analyzed (Participants) | 80
  Duration of illness: 10 to < 20 years | 20
  Duration of illness: > 20 years: number analyzed (Participants) | 48
  Duration of illness: > 20 years | 15
  Smoking history: Absent: number analyzed (Participants) | 188
  Smoking history: Absent | 39
  Smoking history: Present: number analyzed (Participants) | 111
  Smoking history: Present | 35
  Complications: Absent: number analyzed (Participants) | 165
  Complications: Absent | 39
  Complications: Present: number analyzed (Participants) | 231
  Complications: Present | 62
  Complications-renal disorder: Absent: number analyzed (Participants) | 382
  Complications-renal disorder: Absent | 95
  Complications-renal disorder: Present: number analyzed (Participants) | 14
  Complications-renal disorder: Present | 6
  Complications-cardiovascular disorder: Absent: number analyzed (Participants) | 333
  Complications-cardiovascular disorder: Absent | 86
  Complications-cardiovascular disorder: Present: number analyzed (Participants) | 63
  Complications-cardiovascular disorder: Present | 15
  Complications-liver disorder: Absent: number analyzed (Participants) | 366
  Complications-liver disorder: Absent | 95
  Complications-liver disorder: Present: number analyzed (Participants) | 30
  Complications-liver disorder: Present | 6
  Complications-blood disorder: Absent: number analyzed (Participants) | 385
  Complications-blood disorder: Absent | 97
  Complications-blood disorder: Present: number analyzed (Participants) | 11
  Complications-blood disorder: Present | 4
  Complications-respiratory disorder: Absent: number analyzed (Participants) | 372
  Complications-respiratory disorder: Absent | 94
  Complications-respiratory disorder: Present: number analyzed (Participants) | 24
  Complications-respiratory disorder: Present | 7
  Complications-diabetes mellitus: Absent: number analyzed (Participants) | 370
  Complications-diabetes mellitus: Absent | 94
  Complications-diabetes mellitus: Present: number analyzed (Participants) | 26
  Complications-diabetes mellitus: Present | 7
  Complications-uveitis: Absent: number analyzed (Participants) | 355
  Complications-uveitis: Absent | 89
  Complications-uveitis: Present: number analyzed (Participants) | 41
  Complications-uveitis: Present | 12
  Complications-inflammatory bowel disease: Absent: number analyzed (Participants) | 390
  Complications-inflammatory bowel disease: Absent | 100
  Complications-inflammatory bowel disease: Present: number analyzed (Participants) | 6
  Complications-inflammatory bowel disease: Present | 1
  Complications-psoriasis: Absent: number analyzed (Participants) | 391
  Complications-psoriasis: Absent | 100
  Complications-psoriasis: Present: number analyzed (Participants) | 5
  Complications-psoriasis: Present | 1
  Past illnesses: Absent: number analyzed (Participants) | 292
  Past illnesses: Absent | 66
  Past illnesses: Present: number analyzed (Participants) | 94
  Past illnesses: Present | 34
  Allergy history: Absent: number analyzed (Participants) | 336
  Allergy history: Absent | 83
  Allergy history: Present: number analyzed (Participants) | 48
  Allergy history: Present | 12
  Adalimumab self-injection: Absent: number analyzed (Participants) | 131
  Adalimumab self-injection: Absent | 37
  Adalimumab self-injection: Present: number analyzed (Participants) | 265
  Adalimumab self-injection: Present | 64
  Prior medication-NSAIDs: Absent: number analyzed (Participants) | 64
  Prior medication-NSAIDs: Absent | 20
  Prior medication-NSAIDs: Present: number analyzed (Participants) | 332
  Prior medication-NSAIDs: Present | 81
  Prior medication-biological products: Absent: number analyzed (Participants) | 315
  Prior medication-biological products: Absent | 81
  Prior medication-biological products: Present: number analyzed (Participants) | 81
  Prior medication-biological products: Present | 20
  Prior medication-adrenal corticosteroids: Absent: number analyzed (Participants) | 281
  Prior medication-adrenal corticosteroids: Absent | 67
  Prior medication-adrenal corticosteroids: Present: number analyzed (Participants) | 115
  Prior medication-adrenal corticosteroids: Present | 34
  Concomitant drugs: Absent: number analyzed (Participants) | 27
  Concomitant drugs: Absent | 2
  Concomitant drugs: Present: number analyzed (Participants) | 369
  Concomitant drugs: Present | 99
  Concomitant drug-NSAIDs: Absent: number analyzed (Participants) | 127
  Concomitant drug-NSAIDs: Absent | 32
  Concomitant drug-NSAIDs: Present: number analyzed (Participants) | 269
  Concomitant drug-NSAIDs: Present | 69
  Concomitant drug-DMARDs: Absent: number analyzed (Participants) | 186
  Concomitant drug-DMARDs: Absent | 42
  Concomitant drug-DMARDs: Present: number analyzed (Participants) | 210
  Concomitant drug-DMARDs: Present | 59
  Concomitant drug-methotrexate: Absent: number analyzed (Participants) | 247
  Concomitant drug-methotrexate: Absent | 57
  Concomitant drug-methotrexate: Present: number analyzed (Participants) | 149
  Concomitant drug-methotrexate: Present | 44
  Concomitant drug-salazosulfapyridine: Absent: number analyzed (Participants) | 306
  Concomitant drug-salazosulfapyridine: Absent | 78
  Concomitant drug-salazosulfapyridine: Present: number analyzed (Participants) | 90
  Concomitant drug-salazosulfapyridine: Present | 23
  Concomitant drug-adrenal corticosteroids: Absent: number analyzed (Participants) | 288
  Concomitant drug-adrenal corticosteroids: Absent | 63
  Concomitant drug-adrenal corticosteroids: Present: number analyzed (Participants) | 108
  Concomitant drug-adrenal corticosteroids: Present | 38
  Concomitant therapy: Absent: number analyzed (Participants) | 378
  Concomitant therapy: Absent | 97
  Concomitant therapy: Present: number analyzed (Participants) | 18
  Concomitant therapy: Present | 4
  Human leukocyte antigen B27 (HLA-B27): Negative: number analyzed (Participants) | 105
  Human leukocyte antigen B27 (HLA-B27): Negative | 28
  Human leukocyte antigen B27 (HLA-B27): Positive: number analyzed (Participants) | 131
  Human leukocyte antigen B27 (HLA-B27): Positive | 37
  BASDAI: < 4: number analyzed (Participants) | 101
  BASDAI: < 4 | 27
  BASDAI: ≥4: number analyzed (Participants) | 191
  BASDAI: ≥4 | 50
Statistical Analysis 1: Comparison: Adalimumab; Age; Test type: Other; p = 0.0328, Mann-Whitney U-test
Statistical Analysis 2: Comparison: Adalimumab; Sex; Test type: Other; p = 0.7128, Fisher Exact
Statistical Analysis 3: Comparison: Adalimumab; Body mass index; Test type: Other; p = 0.0465, Mann-Whitney U-test
Statistical Analysis 4: Comparison: Adalimumab; Duration of illness; Test type: Other; p = 0.8872, Mann-Whitney U-test
Statistical Analysis 5: Comparison: Adalimumab; Smoking history; Test type: Other; p = 0.0388, Fisher Exact
Statistical Analysis 6: Comparison: Adalimumab; Complications; Test type: Other; p = 0.4855, Fisher Exact
Statistical Analysis 7: Comparison: Adalimumab; Complications - Liver disorder; Test type: Other; p = 0.6630, Fisher Exact
Statistical Analysis 8: Comparison: Adalimumab; Complications - Renal disorder; Test type: Other; p = 0.2067, Fisher Exact
Statistical Analysis 9: Comparison: Adalimumab; Complications - Cardiovascular disorder; Test type: Other; p = 0.8749, Fisher Exact
Statistical Analysis 10: Comparison: Adalimumab; Complications - Blood disorder; Test type: Other; p = 0.4820, Fisher Exact
Statistical Analysis 11: Comparison: Adalimumab; Complications - Respiratory disorder; Test type: Other; p = 0.6355, Fisher Exact
Statistical Analysis 12: Comparison: Adalimumab; Complications - Diabetes mellitus; Test type: Other; p = 0.8193, Fisher Exact
Statistical Analysis 13: Comparison: Adalimumab; Complications - Uveitis; Test type: Other; p = 0.5723, Fisher Exact
Statistical Analysis 14: Comparison: Adalimumab; Complications - Inflammatory bowel disease; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 15: Comparison: Adalimumab; Complications - Psoriasis; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 16: Comparison: Adalimumab; Past Illnesses; Test type: Other; p = 0.0144, Fisher Exact
Statistical Analysis 17: Comparison: Adalimumab; Allergy history; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 18: Comparison: Adalimumab; Adalimumab self-injection status; Test type: Other; p = 0.3928, Fisher Exact
Statistical Analysis 19: Comparison: Adalimumab; Prior medications - NSAIDs; Test type: Other; p = 0.2735, Fisher Exact
Statistical Analysis 20: Comparison: Adalimumab; Prior medications - Biological products; Test type: Other; p = 0.8875, Fisher Exact
Statistical Analysis 21: Comparison: Adalimumab; Prior medications - Adrenal corticosteroids; Test type: Other; p = 0.2540, Fisher Exact
Statistical Analysis 22: Comparison: Adalimumab; Concomitant drugs; Test type: Other; p = 0.0226, Fisher Exact
Statistical Analysis 23: Comparison: Adalimumab; Concomitant drug: NSAIDs; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 24: Comparison: Adalimumab; Concomitant drugs - DMARDs; Test type: Other; p = 0.2481, Fisher Exact
Statistical Analysis 25: Comparison: Adalimumab; Concomitant drugs - Methotrexate; Test type: Other; p = 0.1558, Fisher Exact
Statistical Analysis 26: Comparison: Adalimumab; Concomitant drugs - salazosulfapyridine; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 27: Comparison: Adalimumab; Concomitant drugs - Adrenal corticosteroids; Test type: Other; p = 0.0094, Fisher Exact
Statistical Analysis 28: Comparison: Adalimumab; Concomitant therapy; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 29: Comparison: Adalimumab; Human leukocyte antigen B27 (HLA-B27) test result; Test type: Other; p = 0.8836, Fisher Exact
Statistical Analysis 30: Comparison: Adalimumab; BASDAI at start of treatment; Test type: Other; p = 1.0000, Fisher Exact

3. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage.
Time Frame: 24 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 396
Participants
  Any adverse event | 125
  Serious adverse events | 17

4. Primary Outcome: Number of Participants With Self-injection Errors
Time Frame: 24 weeks
Population: Participants in the safety analysis set who self-injected adalimumab
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 265
Participants | 1

5. Secondary Outcome: Number of Participants With Markedly Improved or Improved Rating
Description: Participants were evaluated for improvement at weeks 12 and 24 of treatment or discontinuation of treatment or participation in the survey based on the clinical course from baseline using the following scale:
  1. Markedly improved, 2. Improved, 3.Not improved, 5. Not assessable
Time Frame: Weeks 12, 24, and at the last visit
Population: Efficacy analysis population; participants with available data at each timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 374
Participants
  12 weeks: number analyzed (Participants) | 287
  12 weeks | 257
  24 weeks: number analyzed (Participants) | 321
  24 weeks | 292
  Last observation | 333

6. Secondary Outcome: Percentage of Participants With Markedly Improved or Improved Rating at Last Visit by Baseline Factors
Description: as for outcome 5
Time Frame: 24 weeks (or last visit if earlier)
Population: Efficacy analysis set; results are only included for participants with non-missing data for each baseline characteristic.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 374
Participants
  Age: 15 to < 65 years: number analyzed (Participants) | 324
  Age: 15 to < 65 years | 291
  Age: ≥ 65 years: number analyzed (Participants) | 50
  Age: ≥ 65 years | 42
  Sex: Male: number analyzed (Participants) | 255
  Sex: Male | 232
  Sex: Female: number analyzed (Participants) | 119
  Sex: Female | 101
  Body Mass Index: < 18.5 kg/m²: number analyzed (Participants) | 31
  Body Mass Index: < 18.5 kg/m² | 25
  Body Mass Index: 18.5 - < 25 kg/m²: number analyzed (Participants) | 158
  Body Mass Index: 18.5 - < 25 kg/m² | 146
  Body Mass Index: 25 - 30 kg/m²: number analyzed (Participants) | 56
  Body Mass Index: 25 - 30 kg/m² | 51
  Body Mass Index: ≥ 30 kg/m²: number analyzed (Participants) | 25
  Body Mass Index: ≥ 30 kg/m² | 20
  Duration of illness: < 5 years: number analyzed (Participants) | 125
  Duration of illness: < 5 years | 113
  Duration of illness: 5 to < 10 years: number analyzed (Participants) | 77
  Duration of illness: 5 to < 10 years | 69
  Duration of illness: 10 to < 20 years: number analyzed (Participants) | 77
  Duration of illness: 10 to < 20 years | 64
  Duration of illness: > 20 years: number analyzed (Participants) | 43
  Duration of illness: > 20 years | 40
  Smoking history: Absent: number analyzed (Participants) | 182
  Smoking history: Absent | 162
  Smoking history: Present: number analyzed (Participants) | 107
  Smoking history: Present | 98
  Complications: Absent: number analyzed (Participants) | 154
  Complications: Absent | 139
  Complications: Present: number analyzed (Participants) | 220
  Complications: Present | 194
  Complications-renal disorder: Absent: number analyzed (Participants) | 360
  Complications-renal disorder: Absent | 321
  Complications-renal disorder: Present: number analyzed (Participants) | 14
  Complications-renal disorder: Present | 12
  Complications-cardiovascular disorder: Absent: number analyzed (Participants) | 314
  Complications-cardiovascular disorder: Absent | 281
  Complications-cardiovascular disorder: Present: number analyzed (Participants) | 60
  Complications-cardiovascular disorder: Present | 52
  Complications-liver disorder: Absent: number analyzed (Participants) | 345
  Complications-liver disorder: Absent | 308
  Complications-liver disorder: Present: number analyzed (Participants) | 29
  Complications-liver disorder: Present | 25
  Complications-blood disorder: Absent: number analyzed (Participants) | 364
  Complications-blood disorder: Absent | 324
  Complications-blood disorder: Present: number analyzed (Participants) | 10
  Complications-blood disorder: Present | 9
  Complications-respiratory disorder: Absent: number analyzed (Participants) | 350
  Complications-respiratory disorder: Absent | 312
  Complications-respiratory disorder: Present: number analyzed (Participants) | 24
  Complications-respiratory disorder: Present | 21
  Complications-diabetes mellitus: Absent: number analyzed (Participants) | 349
  Complications-diabetes mellitus: Absent | 314
  Complications-diabetes mellitus: Present: number analyzed (Participants) | 25
  Complications-diabetes mellitus: Present | 19
  Complications-uveitis: Absent: number analyzed (Participants) | 336
  Complications-uveitis: Absent | 298
  Complications-uveitis: Present: number analyzed (Participants) | 38
  Complications-uveitis: Present | 35
  Complications-inflammatory bowel disease: Absent: number analyzed (Participants) | 369
  Complications-inflammatory bowel disease: Absent | 328
  Complications-inflammatory bowel disease: Present: number analyzed (Participants) | 5
  Complications-inflammatory bowel disease: Present | 5
  Complications-psoriasis: Absent: number analyzed (Participants) | 369
  Complications-psoriasis: Absent | 328
  Complications-psoriasis: Present: number analyzed (Participants) | 5
  Complications-psoriasis: Present | 5
  Past illnesses: Absent: number analyzed (Participants) | 277
  Past illnesses: Absent | 249
  Past illnesses: Present: number analyzed (Participants) | 88
  Past illnesses: Present | 76
  Allergy history: Absent: number analyzed (Participants) | 318
  Allergy history: Absent | 284
  Allergy history: Present: number analyzed (Participants) | 45
  Allergy history: Present | 39
  Adalimumab self-injection: Absent: number analyzed (Participants) | 120
  Adalimumab self-injection: Absent | 101
  Adalimumab self-injection: Present: number analyzed (Participants) | 254
  Adalimumab self-injection: Present | 232
  Prior medication-NSAIDs: Absent: number analyzed (Participants) | 58
  Prior medication-NSAIDs: Absent | 51
  Prior medication-NSAIDs: Present: number analyzed (Participants) | 316
  Prior medication-NSAIDs: Present | 282
  Prior medication-biological products: Absent: number analyzed (Participants) | 301
  Prior medication-biological products: Absent | 272
  Prior medication-biological products: Present: number analyzed (Participants) | 73
  Prior medication-biological products: Present | 61
  Prior medication-adrenal corticosteroids: Absent: number analyzed (Participants) | 263
  Prior medication-adrenal corticosteroids: Absent | 237
  Prior medication-adrenal corticosteroids: Present: number analyzed (Participants) | 111
  Prior medication-adrenal corticosteroids: Present | 96
  Concomitant drugs: Absent: number analyzed (Participants) | 24
  Concomitant drugs: Absent | 22
  Concomitant drugs: Present: number analyzed (Participants) | 350
  Concomitant drugs: Present | 311
  Concomitant drug-NSAIDs: Absent: number analyzed (Participants) | 117
  Concomitant drug-NSAIDs: Absent | 104
  Concomitant drug-NSAIDs: Present: number analyzed (Participants) | 257
  Concomitant drug-NSAIDs: Present | 229
  Concomitant drug-DMARDs: Absent: number analyzed (Participants) | 177
  Concomitant drug-DMARDs: Absent | 157
  Concomitant drug-DMARDs: Present: number analyzed (Participants) | 197
  Concomitant drug-DMARDs: Present | 176
  Concomitant drug-methotrexate: Absent: number analyzed (Participants) | 232
  Concomitant drug-methotrexate: Absent | 202
  Concomitant drug-methotrexate: Present: number analyzed (Participants) | 142
  Concomitant drug-methotrexate: Present | 131
  Concomitant drug-salazosulfapyridine: Absent: number analyzed (Participants) | 291
  Concomitant drug-salazosulfapyridine: Absent | 262
  Concomitant drug-salazosulfapyridine: Present: number analyzed (Participants) | 83
  Concomitant drug-salazosulfapyridine: Present | 71
  Concomitant drug-adrenal corticosteroids: Absent: number analyzed (Participants) | 270
  Concomitant drug-adrenal corticosteroids: Absent | 245
  Concomitant drug-adrenal corticosteroids: Present: number analyzed (Participants) | 104
  Concomitant drug-adrenal corticosteroids: Present | 88
  Concomitant therapy: Absent: number analyzed (Participants) | 356
  Concomitant therapy: Absent | 320
  Concomitant therapy: Present: number analyzed (Participants) | 18
  Concomitant therapy: Present | 13
  Human leukocyte antigen B27 (HLA-B27): Negative: number analyzed (Participants) | 98
  Human leukocyte antigen B27 (HLA-B27): Negative | 83
  Human leukocyte antigen B27 (HLA-B27): Positive: number analyzed (Participants) | 128
  Human leukocyte antigen B27 (HLA-B27): Positive | 121
  BASDAI: < 4: number analyzed (Participants) | 99
  BASDAI: < 4 | 87
  BASDAI: ≥4: number analyzed (Participants) | 184
  BASDAI: ≥4 | 162

7. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) assesses disease activity by asking the participant to answer 6 questions (each on a 10 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For 5 questions (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10 where lower scores indicate less disease activity.
Time Frame: Baseline and weeks 12 and 24
Population: Efficacy analysis population with available BASDAI data at baseline and each timepoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 216
units on a scale
  12 weeks: number analyzed (Participants) | 181
  12 weeks | -1.9 (2.2)
  24 weeks: number analyzed (Participants) | 143
  24 weeks | -2.0 (2.6)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/396
Serious Adverse Events (participants affected / at risk) | 17/396
Other Adverse Events (participants affected / at risk) | 113/396
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=396)
Bronchitis (Infections and infestations) | 2
Impetigo (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaphylactic shock (Immune system disorders) | 1
Myelopathy (Nervous system disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=396)
Bronchitis (Infections and infestations) | 3
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Herpes zoster (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Chlamydial infection (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 2
Tonsillitis bacterial (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypogammaglobulinaemia (Immune system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Anxiety (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Uveitis (Eye disorders) | 2
Vision blurred (Eye disorders) | 1
External ear inflammation (Ear and labyrinth disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Enterocolitis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 1
Swollen tongue (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 12
Hepatic steatosis (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 9
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Lactation disorder (Reproductive system and breast disorders) | 1
Injection site erythema (General disorders) | 4
Injection site pain (General disorders) | 1
Injection site pruritus (General disorders) | 1
Injection site rash (General disorders) | 1
Injection site reaction (General disorders) | 4
Malaise (General disorders) | 3
Thirst (General disorders) | 1
Injection site swelling (General disorders) | 1
Injection site eczema (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 1
Blood urea increased (Investigations) | 2
C-reactive protein increased (Investigations) | 5
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Liver function test abnormal (Investigations) | 3
Lymphocyte count decreased (Investigations) | 4
Lymphocyte count increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Neutrophil count increased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 2
White blood cell count increased (Investigations) | 2
Platelet count increased (Investigations) | 1
Blood beta-D-glucan increased (Investigations) | 1
Blood beta-D-glucan abnormal (Investigations) | 1
Transaminases increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 4
Liver function test increased (Investigations) | 2
Contusion (Injury, poisoning and procedural complications) | 3
Nasopharyngitis (Infections and infestations) | 12
Ophthalmic herpes zoster (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT01329380/Prot_SAP_000.pdf